CLINICAL TRIAL: NCT07251322
Title: Relationship Between Frailty and Gut Microbiota in Older Adults: Relevance for a Healthy Aging Education Program
Brief Title: Relationship Between Frailty and Gut Microbiota in Older Adults: An Educational Program for Healthy Aging
Acronym: FRAGBIOTA
Status: Completed | Type: Observational
Sponsor: University of Cadiz (Other)
Collaborators: Fundación ASISA (Unknown)
Responsible Party: Sponsor
Other Study IDs: FRAGBIOTA
Record Dates: First submitted 2025-09-26; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Frailty; Microbiota
Keywords: gut microbiota; older adults; educational program
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults who participated in an educational intervention program called FRAGSALUD: Participants who, after taking part in an educational intervention of a project called FRAGSALUD, either were considered as responders or non-responders to the intervention, measured if they could reduced their levels of Fried's frailty criteria.
  Interventions: Other: Fecal sample collection

INTERVENTIONS:
Other: Fecal sample collection — Fecal samples were collected by the participants themselves at home, who were instructed to collect a small stool sample either on the morning of the delivery day or the evening of the previous day. For home sample collection, participants were provided with a fecal sample collection kit that included a hermetically sealed sterile container, a fecal sample stabilizer (reference SC0012, Canvax brand), gloves, and a small spoon. Participants were instructed to collect a small fecal sample using the spoon and place it into the container, mixing it by shaking to combine it with the stabilizer.

SUMMARY:
The main objective of this pre-experimental study is to describe the relationship between gut microbiota and changes in the degree of frailty in older adults who participated in an educational program. More specifically, the study aims to: determine the gut microbiota profile of community-dwelling older adults, both robust and frail; analyze the effect of a 12-month educational program on gut microbiota; examine the association of gut microbiota with physical function, functional dependency, and physical activity in frail or pre-frail older adults who received the program; investigate its relationship with the risk of malnutrition; relate the gut microbiota profile to quality of life, depressive symptoms, and social support; and, finally, associate gut microbiota with cognitive frailty and sleep quality in this group of older adults who participated in the health promotion educational intervention.

DETAILED DESCRIPTION:
This non-randomized pre-experimental study was conducted in the province of Cádiz, Spain. A total of 14 older adults participated, all of whom had previously taken part in the intervention group of the randomized experimental project called Fragsalud, which aimed to improve frailty through educational sessions. During that project, frailty was assessed using the Fried criteria, and physical condition, physical activity, and sleep were evaluated through accelerometry, as well as questionnaires on nutritional habits, depressive symptoms, social support, instrumental and basic activities of daily living, quality of life, cognition, and sleep, at the beginning of the study, at 6 months, and at the end of the study at 12 months. For the Fragbiota project, once Fragsalud was completed, participants were analyzed based on whether or not they responded to the educational intervention. That is, the gut microbiota of those subjects who, after 12 months, had reduced the Fried frailty criteria was compared with those who, despite receiving the educational intervention, had maintained the same Fried levels or had worsened. Furthermore, this gut microbiota was related to the secondary variables previously assessed in the Fragsalud project. This study complied with biomedical ethical guidelines, including Good Clinical Practice (CPMP/ICH/135/95), the Oviedo Convention, the Universal Declaration of Human Rights, CIOMS/WHO ethical guidelines, and the Declaration of Helsinki, ensuring the dignity, rights, and safety of participants. Additionally, participants provided informed consent after receiving detailed explanations, both in writing and verbally, regarding the objectives, procedures, and risks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age who present frailty or pre-frailty, assessed using the Fried criteria adapted to the Spanish population
* Patients belonging to the Clinical Management Units participating in the study and who will remain in them for the 12 months of the study
* Patients who are able to attend the Health Center alone or accompanied

Exclusion Criteria:

* COPD stage III or IV, unstable angina, uncontrolled congestive heart failure, or unstable arrhythmia
* Patients who cannot walk independently or with assistive devices, such as bedridden individuals
* Patients in nursing homes
* Patients with severe cognitive impairment
* Patients who do not understand Spanish or English
* Patients with allergies to plastic or metal

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A cohort of participants of the FRAGSALUD project (older adults with at least one Fried's frailty criterion), that will be divided into to responders (if they reduced their levels of frailty) and non-responders (if they did not reduced their levels of frailty) after the FRAGSALUD intervention (an educactional program of four sessions and six telephone calls)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Gut microbiota | At 12 months after the completion of the study
  Fecal samples will be collected by the participants themselves at home. For the determination of gut microbiota, the following steps will be carried out:
  DNA Extraction: DNA will be extracted using the QIAamp DNA Stool Mini Kit (QIAGEN, Barcelona, Spain).
  Sequencing: Polymerase Chain Reaction (PCR) will be used to amplify the extracted DNA with primers targeting the hypervariable V3 and V4 regions of the bacterial 16S rRNA gene, using the following primers: forward 16S Amplicon PCR primer: 5'TCGTCGGCAGCGTCAGATGTGTATAAGAGACAGCCTACGGGNGGCWGCAG, and reverse 16S Amplicon PCR primer: 5'GTCTCGTGGGCTCGGAGATGTGTATAAGAGACAGGACTACHVGGGTATCTAATCC.
  Bioinformatic Analysis: Illumina bcl2fastq2 v2.20 software will be used to demultiplex the raw sequences, and the raw data will be imported into the open-source QIIME 2 2020.8 software.
  Functional Profile Determination: PICRUSt2 will be used to predict potential functional profiles for the sequenced samples.

SECONDARY OUTCOMES:
Frailty Index | Day one and at 12 months after the completion of the study
  Through the Fried questionnaire, which includes five domains: i) unintentional weight loss, ii) self-reported exhaustion and fatigue, iii) low weekly physical activity measured using the short version of the Minnesota Leisure Time Physical Activity Questionnaire, iv) gait speed over 4.57 meters, and v) low grip strength measured with a hand-held dynamometer.
Functional capacity or physical performance | Day one and at 12 months after the completion of the study
  Using the Short Physical Performance Battery (SPPB), balance was assessed (with the feet together, semi-tandem, and tandem tests), gait speed was measured (with the 4-meter walking test), and lower body strength was evaluated (with the five-times chair stand test).
Functional dependence | Day one and at 12 months after the completion of the study
  Functional dependence was assessed using the Barthel Index, which is a reliable and validated tool designed to evaluate an individual's ability to perform ten Activities of Daily Living. These activities include feeding, transferring from a chair to the bed, bathing, dressing, grooming, bowel control, bladder control, using the toilet, walking, and climbing stairs. Additionally, the Lawton and Brody scale was applied, which is a reliable and validated tool used to assess Instrumental Activities of Daily Living, covering eight domains: use of the telephone, transportation, medication management, financial transactions, meal preparation, shopping, household maintenance, and laundry.
Physical activity and sleep patterns | Day one and at 12 months after the completion of the study
  Measured using wrist-worn accelerometers (GENEActiv, ActivInsights Ltd., Kimbolton, UK), which participants wore for at least six consecutive days. The accelerometers were set to 60 Hz, and raw data were downloaded using GENEActiv software version 3.3. All raw data files were analyzed on the servers of the University of Málaga using the open-source R package GGIR, version 2.7-0. This R package auto-calibrated the data according to local gravity and calculated the Euclidean Norm Minus One (ENMO) for accelerations to minimize sensor calibration error.
Subjective sleep | Day one and at 12 months after the completion of the study
  Using the Pittsburgh Sleep Quality Index, which has been validated in this population, the questionnaire includes 19 items assessing seven distinct dimensions of sleep. These dimensions include subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, use of sleep medication, and daytime dysfunction.
Quality of life assessment | Day one and at 12 months after the completion of the study
  The EuroQoL 5-Dimension 5-Level (EQ-5D-5L) was used to assess health-related quality of life in the older participants. It consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), with participants rating each dimension on a five-point scale from 1 (no problems) to 5 (extreme problems). These ratings were combined into a five-digit number representing their health state. After generating 3,125 possible health states, a formula was used to convert them into a single health index ranging from 0 to 1, with 1 representing the maximum achievable score. In addition, the questionnaire included a Visual Analog Scale (VAS) to assess self-reported health levels. The VAS consisted of a scale from 0 (representing the worst imaginable health state) to 100 (representing the best imaginable health state), and participants were asked to indicate the score that best represented their health on the day of the assessment.
Depressive symptoms | Day one and at 12 months after the completion of the study
  Through the 15-item Yesavage Geriatric Depression Scale (GDS-15), a validated assessment tool for depression in older adults. The GDS-15 uses a binary response format (yes or no) and evaluates only the cognitive symptoms of a major depressive episode experienced during the past 15 days, excluding somatic depressive symptoms such as sleep difficulties, changes in appetite, lack of concentration, and fatigue.
Social support | Day one and at 12 months after the completion of the study
  Through the Duke-UNC Functional Social Support Questionnaire (Duke-UNC-11), which has been validated in the Spanish population.
Cognitive function assessment | Day one and at 12 months after the completion of the study
  The cognitive status of the participants was assessed using the Portable Short Portable Mental Status Questionnaire (SPMSQ), which has demonstrated good validity and reliability in the Spanish population. This test is widely used due to its brevity and ease of administration, making it a rapid screening tool. It consists of 10 questions that evaluate short- and long-term memory, orientation, and the ability to perform serial mathematical tasks.
Risk of malnutrition | Day one and at 12 months after the completion of the study
  Through the Mini-Nutritional Assessment (MNA). This evaluation includes questions related to various aspects such as lifestyle, medication, mobility, number of meals, food and fluid intake, independence in eating, and self-perception of health and nutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Casals Vázquez, Principal Investigator — University of Cádiz; Juan Corral Pérez, Principal Investigator — University of Cádiz
Locations (1):
- Facultad de Ciencias de la Educación, Puerto Real, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Undecided